CLINICAL TRIAL: NCT00258895
Title: Safety and Immunogenicity of DAPTACEL® Administered as a 5th Dose in 4 to 6-Year-Old Children Previously Immunized With DAPTACEL® or Pentacel®
Brief Title: Safety and Immunogenicity of DAPTACEL® as 5th Dose in Children 4 to 6 Years Old After 4 Doses of Pentacel™ or DAPTACEL®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P3T11
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: DAPTACEL®; Pentacel™; Diphtheria; Tetanus; Pertussis; Whooping cough; Acellular Pertussis Vaccine Adsorbed
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines

ARMS (2):
- DAPTACEL Primed (Experimental): Participants received Daptacel in Study P3T06.
  Interventions: Biological: DAPTACEL®: DTaP
- Pentacel Primed (Experimental): Participants received Pentacel in Study P3T06
  Interventions: Biological: DAPTACEL®: DTaP

INTERVENTIONS:
Biological: DAPTACEL®: DTaP — 0.5 mL, Intramuscular
  Other Names: DAPTACEL®
  Arms: DAPTACEL Primed
Biological: DAPTACEL®: DTaP — 0.5 mL, Intramuscular
  Other Names: DAPTACEL®
  Arms: Pentacel Primed

SUMMARY:
Primary Objectives:

1. To present the safety profile after a 5th dose of DAPTACEL® in children 4 to 6 years of age who have previously received 4 doses of DAPTACEL® or Pentacel™.
2. To present the pre-Dose 5 and post-Dose 5 antibody responses to the antigens in DAPTACEL® in children 4 to 6 years of age who have previously received 4 doses of DAPTACEL® or Pentacel™.

Observational Objectives:

1. To compare under equivalence criteria the pre-Dose 5 and post-Dose 5 antibody responses to the antigens in DAPTACEL® in children 4 to 6 years of age who have previously received 4 doses of DAPTACEL® or Pentacel™.
2. To present the pre-vaccination anti-poliovirus GMTs and seroprotection rates.
3. To present the post-vaccination anti-poliovirus GMTs and seroprotection rates among subjects receiving a 4th dose of IPV concurrently with the 5th dose of DAPTACEL and a 2nd dose of MMR.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 4 and < 7 years from date of birth at the time of study vaccination
* Signed and dated Investigational Review Board (IRB)-approved informed consent from a parent or legally authorized representative. Signed and dated IRB-approved assent from subject if required by IRB
* Judged to be in good health on the basis of reported medical history and physical examination
* Able and willing to attend the scheduled visits and to comply with the study procedures
* Has documented complete infant series and the 4th dose of DAPTACEL® or Pentacel™ in Study P3T06 (i.e., 4 previous administrations of DAPTACEL® or Pentacel™).

Exclusion Criteria:

* Received a 5th dose of DTaP-containing vaccine
* a. For subjects in the DAPTACEL® arm: Received a 4th dose of Inactivated Poliovirus Vaccine (IPV) vaccine and/or a 2nd dose of Measles, Mumps, and Rubella (MMR) vaccine scheduled at 4 to 6 years of age.

  b. For subjects in the Pentacel™ arm: Received a 2nd dose of MMR vaccine scheduled at 4 to 6 years of age
* Severe hypersensitivity to any component of the vaccine such as an anaphylactic reaction observed following a previous vaccination
* Serious underlying chronic disease, including, but not limited to:·Diabetes mellitus; malignancy; cardiopulmonary disease; renal, endocrinologic, or hepatic dysfunction; or hematologic disorder·Unstable or evolving neurologic disorders that may predispose the subject to seizures or neurologic deterioration. These may include progressive neurologic disorders (e.g., infantile spasms, uncontrolled progressive encephalopathy) and encephalopathy within 7 days following previous vaccination
* Known or suspected primary or acquired disease of the immune system
* Administration of immune globulin, other blood products within the last 3 months, injected or oral corticosteroids or other immunomodulator therapy within 6 weeks prior to study vaccination. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than 1 course within the last 2 weeks prior to enrollment
* Had allergy shots started or had changes in regimen or dosing of allergy shots within 4 weeks prior to study vaccination
* Receipt of any other vaccine within 30 days prior to study vaccination, or planning to receive another vaccine within 30 days before the Visit 2 blood draw (if applicable)
* Any other condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine
* Enrolled in another vaccine trial
* Personal history of physician-diagnosed or laboratory-confirmed pertussis disease within the past 30 months
* Known or suspected allergy to any of the vaccines or vaccine components intended for use in this study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 649 (Actual)
Dates: Start 2005-03; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (21):
- United States (21):
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Centennial, Colorado
  - Norwich, Connecticut
  - Marietta, Georgia
  - Bardstown, Kentucky
  - Bossier City, Louisiana
  - Rochester, New York
  - Pembroke, North Carolina
  - Sylva, North Carolina
  - Norristown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Kingsport, Tennessee
  - Fort Worth, Texas
  - San Antonio, Texas
  - Provo, Utah
  - Spokane, Washington
  - La Crosse, Wisconsin
  - Marshfield, Wisconsin

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 30 March 2005 to 02 March 2006 at 22 US sites.
Pre-assignment Details: A total of 649 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- DAPTACEL®-Primed: Participants received Daptacel in Study P3T06; and a fifth dose of DAPTACEL® vaccine concurrently with a fourth dose of inactivated poliovirus vaccine in this study.
- Pentacel®-Primed: Participants received Pentacel in Study P3T06, received a fifth dose of DAPTACEL® vaccine after 4 doses of Pentacel® vaccine in this study.
Period: Overall Study
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed
Started | 487 | 162
Completed | 477 | 159
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed | Total
Number analyzed (Participants) | 487 | 162 | 649
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 487 | 162 | 649
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.1 (0.14) | 4.1 (0.16) | 4.1 (0.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 83 | 327
  Male | 243 | 79 | 322
Region of Enrollment [Number; unit: participants]
  United States | 487 | 162 | 649

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Local or Systemic Reactions Post-Dose 5 of DAPTACEL® Vaccination
Time Frame: 0 to 7 days Post-Dose 5
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed
Number analyzed (Participants) | 485 | 162
Percentage of Participants
  Any Solicited Local Reaction - Dose 5 | 75 | 70
  Any Redness (> 5 mm) | 36 | 24
  Grade 3 Redness (> 50 mm) | 16 | 9
  Any Swelling (> 5 mm) | 24 | 14
  Grade 3 Swelling (> 50 mm) | 8 | 1
  Any Tenderness | 62 | 55
  Grade 3 Tenderness (Incapacitating) | 2 | 0
  Any Change in Limb Circumference (> 5 mm) | 39 | 32
  Grade 3 Change in Limb Circumference (> 40 mm) | 2 | 0
  Any Functional Impairment | 20 | 12
  Grade 3 Functional Impairment (Incapacitating) | 0 | 0
  Any Solicited Systemic Reaction - Dose 5 | 55 | 45
  Any Fever (≥ 38.0 ºC) | 8 | 6
  Grade 3 Fever (> 39.5 ºC) | 0 | 1
  Any Irritability | 36 | 28
  Grade 3 Irritability (Incapacitating) | 0 | 0
  Any Crying | 15 | 11
  Grade 3 Crying (Incapacitating) | 0 | 0
  Any Lethargy | 22 | 17
  Grade 3 Lethargy (Incapacitating) | 1 | 1
  Any Anorexia | 16 | 14
  Grade 3 Anorexia (skipped 2 meals) | 1 | 1
  Any Vomiting (per 24 hours) | 4 | 4
  Grade 3 Vomiting (≥ 3 episodes) | 1 | 0
  Any Diarrhea (per 24 hours) | 8 | 6
  Grade 3 Diarrhea (> 5 diarrhea stools) | 0 | 0
  Any Rash | 10 | 5

2. Primary Outcome: Percentage of Participants With Anti-Pertussis 4-Fold Rises Post-Dose 5 of DAPTACEL® Vaccination
Description: Anti-Pertussis (anti-Pertussis, anti-Filamentous Haemagglutinin, anti-Fimbriae, and anti-Pertactin) Fold-rise is calculated as post-Dose 5/pre-Dose 5 titer.
Time Frame: Day 28 to 48 Post-dose 5
Population: The anti-Pertussis 4-fold rises were evaluated in the per-protocol immunology population.
Measure: Number; unit: Percentage of Participants
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed
Number analyzed (Participants) | 251 | 80
Percentage of Participants
  Anti-Pertussis (EU/mL) | 92 | 98
  Anti-Filamentous Haemagglutinin (EU/mL) | 89 | 89
  Anti-Fimbriae Types 2 and 3 (EU/mL) | 90 | 96
  Anti-Pertactin (EU/mL) | 94 | 95

3. Primary Outcome: Percentage of Participants With Anti-Pertussis Booster Response Post-Dose 5 of DAPTACEL® Vaccination
Description: Booster response calculation: If pre-Dose 5 titer < 4x limit of quantitation (LOQ) a 4-fold rise of post-Dose 5/pre-Dose 5. If pre-Dose 5 titer ≥ 4x LOQ a 2-fold rise of post-Dose 5/pre-Dose 5.
Time Frame: Day 28 to 48 Post-Dose 5
Population: The anti-pertussis booster response was assessed in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed
Number analyzed (Participants) | 251 | 80
Percentage of Participants
  Anti-Pertussis (EU/mL) | 96 | 99
  Anti-Fillamentous Haemagglutinin (EU/mL) | 93 | 96
  Anti-Fimbriae Types 2 and 3 (EU/mL) | 96 | 99
  Anti-Pertactin (EU/mL) | 97 | 96

4. Primary Outcome: Percentage of Participants With Anti-Diphtheria and Anti-Tetanus Toxoids Responses Pre- and Post-Dose 5 of DAPTACEL® Vaccination.
Time Frame: Day 0 and between Days 28-48 Post-dose 5
Population: Antibody responses were assessed for each of the antigens in DAPTACEL vaccine in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of Participants
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed
Number analyzed (Participants) | 251 | 81
Percentage of Participants
  Anti-Diphtheria (IU/mL) ≥ 0.01 Pre-dose 5 | 99 | 99
  Anti-Diphtheria (IU/mL) ≥ 0.1 Pre-dose 5 | 47 | 50
  Anti-Diptheria (IU/mL) ≥ 1.0 Pre-dose 5 | 1 | 1
  Anti-Diphtheria (IU/mL) ≥ 0.1 Post-dose 5 | 100 | 100
  Anti-Diphtheria (IU/mL) ≥ 1.0 Post-dose 5 | 100 | 100
  Anti-Tetanus (IU/mL) ≥ 0.01 Pre-dose 5 | 100 | 99
  Anti-Tetanus (IU/mL) ≥ 0.1 Pre-dose 5 | 85 | 82
  Anti-Tetanus (IU/mL) ≥ 1.0 Pre-dose 5 | 20 | 12
  Anti-Tetanus (IU/mL) ≥ 0.1 Post-dose 5 | 100 | 100
  Anti-Tetanus (IU/mL) ≥ 1.0 Post-dose 5 | 99 | 98

5. Primary Outcome: Geometric Mean Titers (GMTs) of Anti-Pertussis, Anti-Diphtheria, and Anti-Tetanus Toxoids Pre- and Post-dose 5 of DAPTACEL® Vaccination
Time Frame: Day 0 and between Days 28-48 post-dose 5
Population: GMTs were assessed for each of the antigens in DAPTACEL vaccine in the per-protocol immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: All units
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed
Number analyzed (Participants) | 255 | 81
All units
  Anti-Pertussis (EU/mL) Pre-Dose | 7.67 [6.66 to 8.84] | 9.80 [7.81 to 12.29]
  Anti-Pertussis (EU/mL) Post-Dose | 154.32 [139.58 to 170.62] | 180.77 [150.33 to 217.38]
  Anti-Filamentous Haemagglutinin (EU/mL) Pre-Dose | 5.03 [4.25 to 5.96] | 7.52 [5.45 to 10.39]
  Anti-Filamentous Haemagglutinin (EU/mL) Post-Dose | 82.11 [73.39 to 91.88] | 120.03 [98.10 to 146.86]
  Anti-Fimbriae Types 2 and 3 (EU/mL) Pre-dose | 24.45 [21.22 to 28.16] | 34.50 [27.00 to 44.09]
  Anti-Fimbriae Types 2 and 3 (EU/mL) Post-dose | 450.56 [407.40 to 498.30] | 649.86 [551.73 to 765.45]
  Anti-Pertactin (EU/mL) Pre-dose | 15.62 [13.72 to 17.78] | 9.16 [7.10 to 11.81]
  Anti-Pertactin (EU/mL) Post-dose | 229.59 [207.45 to 254.08] | 148.80 [120.63 to 183.55]
  Anti-Diphtheria (IU/mL) Pre-dose | 0.11 [0.09 to 0.12] | 0.11 [0.08 to 0.14]
  Anti-Diphtheria (IU/mL) Post-dose | 19.59 [17.06 to 22.51] | 22.56 [17.78 to 28.62]
  Anti-Tetanus (IU/mL) Pre-dose | 0.38 [0.33 to 0.43] | 0.27 [0.21 to 0.34]
  Anti-Tetanus (IU/mL) Post-dose | 6.21 [5.59 to 6.89] | 4.47 [3.75 to 5.34]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 6 months post-vaccination.
Arm/Group | DAPTACEL®-Primed | Pentacel®-Primed
Serious Adverse Events (participants affected / at risk) | 5/487 | 3/162
Other Adverse Events (participants affected / at risk) | 62/487 | 55/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPTACEL®-Primed (N=487) | Pentacel®-Primed (N=162)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastroenteritis NOS (Infections and infestations) | 0 (0) | 2 (2)
Otitis media NOS (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture NOS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Staring (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma NOS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DAPTACEL®-Primed (N=487) | Pentacel®-Primed (N=162)
Injection site redness (General disorders) | 36 | 24
Injection site swelling (General disorders) | 24 | 14
Injection site tenderness (General disorders) | 62 | 55
Irritability (Psychiatric disorders) | 36 | 28
Crying (Psychiatric disorders) | 15 | 11
Anorexia (Musculoskeletal and connective tissue disorders) | 16 | 14
Lethargy (Gastrointestinal disorders) | 22 | 17
Otitis media NOS (Infections and infestations) | 24 | 9
Upper respiratory tract infection NOS (Infections and infestations) | 34 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.